CLINICAL TRIAL: NCT00615992
Title: Effect of Spiriva on the Activities of Daily Living Score Recommended in Austrian COPD Guidelines
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 205.398
Record Dates: First submitted 2008-01-24; First posted 2008-02-14 (Estimated); Results first posted 2009-12-24 (Estimated); Last update posted 2016-02-08 (Estimated); Status verified 2016-01

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Tiotropium Bromide

STUDY DESIGN:
Observational Model: Cohort

INTERVENTIONS:
Drug: Tiotropium

SUMMARY:
The primary goal of this post marketing surveillance (PMS) study is to document the efficacy of Tiotropium (Spiriva) to improve physical activity measured by a score that is recommended in national chronic obstructive pulmonary disease (COPD) guidelines for monitoring the course of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspected chronic obstructive pulmonary disease (COPD)
* 3 or more positive answers in COPD questionnaire
* Age over 40 years

Exclusion Criteria:

* Patients with any conditions listed in special precautions, drug interactions, and contraindication of Spiriva in the summary of product characteristics
* Patient treated with Spiriva in the past year
* Patient with history of hypersensitivity to tiotropium bromide, atropine and/or its derivant, i.e. ipratropium, or any component of Spiriva Patient with known narrow-angle glaucoma Patient with known symptomatic prostatic hyperplasia and/or bladder-neck obstruction Patient with known moderate to severe renal impairment (i.e.,creatinine clearance<=50ml/min) Pregnant or nursing women Patient with any significant disease other than COPD which would exclude him/her from participating in the study Patients with any conditions listed in special precautions, drug interactions, and contraindication of Spiriva in Austrian summary of product characteristics

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care
Sampling Method: Probability Sample
Enrollment: 754 (Actual)
Dates: Start 2007-04; Primary Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (73):
- Austria (73):
  - Boehringer Ingelheim Investigational Site, Admont
  - Boehringer Ingelheim Investigational Site, Afritz Am See
  - Boehringer Ingelheim Investigational Site, Altenmarkt
  - Boehringer Ingelheim Investigational Site, Altmünster
  - Boehringer Ingelheim Investigational Site, Bad Gleichenberg
  - Boehringer Ingelheim Investigational Site, Bad Goisern am Hallstättersee
  - Boehringer Ingelheim Investigational Site, Bad Hall
  - Boehringer Ingelheim Investigational Site, Bad Häring
  - Boehringer Ingelheim Investigational Site, Bleiburg
  - Boehringer Ingelheim Investigational Site, Bludenz
  - Boehringer Ingelheim Investigational Site, Brixlegg
  - Boehringer Ingelheim Investigational Site, Drasenhofen
  - Boehringer Ingelheim Investigational Site, Enns
  - Boehringer Ingelheim Investigational Site, Fohnsdorf
  - Boehringer Ingelheim Investigational Site, Gänserndorf
  - Boehringer Ingelheim Investigational Site, Gmunden
  - Boehringer Ingelheim Investigational Site, Grafenstein
  - Boehringer Ingelheim Investigational Site, Graz
  - Boehringer Ingelheim Investigational Site, Grünbach
  - Boehringer Ingelheim Investigational Site, Gunskirchen
  - Boehringer Ingelheim Investigational Site, Gutenstein
  - Boehringer Ingelheim Investigational Site, Haid
  - Boehringer Ingelheim Investigational Site, Hainburg/a.d. Donau
  - Boehringer Ingelheim Investigational Site, Herzogenburg
  - Boehringer Ingelheim Investigational Site, Hürm
  - Boehringer Ingelheim Investigational Site, Innsbruck
  - Boehringer Ingelheim Investigational Site, Jenbach
  - Boehringer Ingelheim Investigational Site, Judenburg
  - Boehringer Ingelheim Investigational Site, Kindberg
  - Boehringer Ingelheim Investigational Site, Kirchberg Wechsel
  - Boehringer Ingelheim Investigational Site, Klagenfurt
  - Boehringer Ingelheim Investigational Site, Klein-Pöchlarn
  - Boehringer Ingelheim Investigational Site, Knittelfeld
  - Boehringer Ingelheim Investigational Site, Königswiesen
  - Boehringer Ingelheim Investigational Site, Kuchl
  - Boehringer Ingelheim Investigational Site, Langenrohr
  - Boehringer Ingelheim Investigational Site, Lebring
  - Boehringer Ingelheim Investigational Site, Leobersdorf
  - Boehringer Ingelheim Investigational Site, Linz
  - Boehringer Ingelheim Investigational Site, Lustenau
  - Boehringer Ingelheim Investigational Site, Mank
  - Boehringer Ingelheim Investigational Site, Mödling
  - Boehringer Ingelheim Investigational Site, Neuberg/Mürz
  - Boehringer Ingelheim Investigational Site, Neumarkt a.W.
  - Boehringer Ingelheim Investigational Site, Neunkirchen
  - Boehringer Ingelheim Investigational Site, Niederhollabrunn
  - Boehringer Ingelheim Investigational Site, Oberschützen
  - Boehringer Ingelheim Investigational Site, Ollersdorf
  - Boehringer Ingelheim Investigational Site, Passail
  - Boehringer Ingelheim Investigational Site, Peesen
  - Boehringer Ingelheim Investigational Site, Pfarrkirchen bei Bad Hall
  - Boehringer Ingelheim Investigational Site, Pichl bei Wels
  - Boehringer Ingelheim Investigational Site, Pischeldorf
  - Boehringer Ingelheim Investigational Site, Rattenberg
  - Boehringer Ingelheim Investigational Site, Saint Johann
  - Boehringer Ingelheim Investigational Site, Saint Stefan O Stainz
  - Boehringer Ingelheim Investigational Site, Saint Veit Glan
  - Boehringer Ingelheim Investigational Site, Salzburg
  - Boehringer Ingelheim Investigational Site, Sankt Valentin
  - Boehringer Ingelheim Investigational Site, Schwechat
  - Boehringer Ingelheim Investigational Site, St.Georgen/Judenburg 12
  - Boehringer Ingelheim Investigational Site, Stainach
  - Boehringer Ingelheim Investigational Site, Stasshof
  - Boehringer Ingelheim Investigational Site, Traismauer
  - Boehringer Ingelheim Investigational Site, Tulln
  - Boehringer Ingelheim Investigational Site, Vienna
  - Boehringer Ingelheim Investigational Site, Vöcklabruck
  - Boehringer Ingelheim Investigational Site, Wallern an der Trattnach
  - Boehringer Ingelheim Investigational Site, Weiz
  - Boehringer Ingelheim Investigational Site, Weißtrach
  - Boehringer Ingelheim Investigational Site, Wilhelmsburg
  - Boehringer Ingelheim Investigational Site, Wolfsberg
  - Boehringer Ingelheim Investigational Site, Wolkersdorf

RESULTS

PARTICIPANT FLOW:
Groups:
- Spiriva® (Tiotropium Bromide): Tiotropium bromide 18μg inhalation capsules once-daily
Period: Overall Study
Arm/Group | Spiriva® (Tiotropium Bromide)
Started | 754
Completed | 687
Not Completed | 67
Not completed — Protocol Violation | 67

BASELINE CHARACTERISTICS:
Arm/Group | Spiriva® (Tiotropium Bromide)
Number analyzed (Participants) | 687
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.0 (12.5)
Sex/Gender, Customized [Number; unit: participants] — 687 eligible for efficacy analysis (complete data set available)
  Throughout this report, the discrepancy between the total number of participants and the numbers analyzed for a certain parameter is due to missing data.
  Number of Participant in this summary is "number of patients used for analysis".
  participants
    Female | 269
    Male | 414
    Missing | 4

OUTCOME MEASURES:

1. Primary Outcome: Activities of Daily Living Score After 3 to 4 Weeks Treatment With Spiriva
Description: The scores are final, not a difference in score. Rating scale scored from 0 (no restrictions in activities) to 4 (severe restrictions)
Time Frame: Protocol-defined treatment period between initiation of therapy with Spiriva and the final visit (21 to 28 days)
Population: The discrepancy between the total number of participants and the numbers analyzed for a certain parameter is due to missing data.
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Spiriva® (Tiotropium Bromide)
Number analyzed (Participants) | 687
points on a scale | 1.1 (0.7)

2. Secondary Outcome: Dyspnea Score After 3 to 4 Weeks Treatment With Spiriva
Description: as for outcome 1
Time Frame: Protocol-defined treatment period between initiation of therapy with Spiriva and the final visit (21 to 28 days)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Spiriva® (Tiotropium Bromide)
Number analyzed (Participants) | 687
points on a scale | 1.1 (0.7)

3. Secondary Outcome: Global Assessment of Efficacy by Patient
Description: Rating scale ranging from very good (best value) to not satisfactory (worst value)
Time Frame: Protocol-defined treatment period between initiation of therapy with Spiriva and the final visit (21 to 28 days)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Spiriva® (Tiotropium Bromide)
Number analyzed (Participants) | 646
Participants
  Very good | 373
  Good | 217
  Satisfactory | 53
  Not satisfactory | 3

4. Secondary Outcome: Global Assessment of Tolerability by Patient
Description: Rating scale ranging from very good (best value) to not satisfactory (worst value)
Time Frame: Protocol-defined treatment period between initiation of therapy with Spiriva and the final visit (21 to 28 days)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Spiriva® (Tiotropium Bromide)
Number analyzed (Participants) | 647
Participants
  Very good | 493
  Good | 142
  Satisfactory | 11
  Not satisfactory | 1

5. Secondary Outcome: Global Assessment of Efficacy by Physician
Description: Rating scale ranging from very good (best value) to not satisfactory (worst value)
Time Frame: Protocol-defined treatment period between initiation of therapy with Spiriva and the final visit (21 to 28 days)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Spiriva® (Tiotropium Bromide)
Number analyzed (Participants) | 648
Participants
  Very good | 407
  Good | 205
  Satisfactory | 36
  Not satisfactory | 0

6. Secondary Outcome: Global Assessment of Tolerability by Physician
Description: Rating scale ranging from very good (best value) to not satisfactory (worst value)
Time Frame: Protocol-defined treatment period between initiation of therapy with Spiriva and the final visit (21 to 28 days)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Spiriva® (Tiotropium Bromide)
Number analyzed (Participants) | 647
Participants
  Very good | 540
  Good | 102
  Satisfactory | 5
  Not satisfactory | 0

ADVERSE EVENTS:
Time Frame: 4 Weeks
Arm/Group | Spiriva® (Tiotropium Bromide)
Serious Adverse Events (participants affected / at risk) | 0/754
Other Adverse Events (participants affected / at risk) | 0/754

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.